CLINICAL TRIAL: NCT03740230
Title: Post-marketing Surveillance to Assess the Safety and Effectiveness of Maviret (Glecaprevir/Pibrentasvir) for Korean Chronic Hepatitis C Genotypes 1 to 6 Patients According to the "Standard for Re-examination of New Drugs"
Brief Title: An Observational Study of Maviret (Glecaprevir/Pibrentasvir) for Korean Chronic Hepatitis C Genotypes 1 to 6 Patients According to the Standard for Re-examination of New Drugs
Acronym: Maviret PMS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-423
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Chronic Hepatitis C; Genotypes; Genotypes 1 to 6; Maviret; Glecaprevir; Pibrentasvir
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hepatitis C: Participants with Hepatitis C Genotypes 1 to 6 receiving Maviret (glecaprevir/pibrentasvir) for 8, 12, or 16 weeks.

SUMMARY:
Post-marketing surveillance study to evaluate the real world safety and effectiveness of Maviret (Glecaprevir/Pibrentasvir) administered under a normal, routine treatment practice by Korean patients with Chronic Hepatitis C Genotypes 1 to 6

DETAILED DESCRIPTION:
Patients with type C hepatitis genotypes 1-6 who had been prescribed Maviret (glecaprevir/pibrentasvir) in accordance with approved local label.

The sample size for this study is due to a requirement by local authorities.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic C hepatitis genotypes 1 to 6.
* Participants prescribed Maviret in accordance with approved local label.

Exclusion Criteria:

- Patients with contraindications to the approved local labels for Maviret.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Hepatitis C Genotypes 1 to 6 receiving Maviret (glecaprevir/pibrentasvir) for 8, 12, or 16 weeks.
Sampling Method: Probability Sample
Enrollment: 3134 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12) | 12 weeks after the last dose of study drug
  SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after end of treatment.

SECONDARY OUTCOMES:
Percentage of Participants With On-treatment Virologic Failure | Up to 30 weeks
  On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or HCV RNA ≥ LLOQ persistently during treatment period.
Percentage of Participants With Post-treatment Relapse | Up to 28 weeks
  Post-treatment relapse defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after the end of treatment among participants who complete treatment and with HCV RNA levels < LLOQ at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (61):
- South Korea (61):
  - SoonChunHyang University CheonAn Hospital /ID# 209996, Cheonan-si, Chungcheongnam-do
  - Hallym University Sacred Heart Hospital /ID# 210809, Anyang, Gyeonggido
  - The Catholic University of Korea, Bucheon St.Mary's Hospital /ID# 216869, Bucheon-si, Gyeonggido
  - Dongguk University Ilsan Hospital /ID# 210609, Goyang, Gyeonggido
  - National health insurance Service ilsanhospital /ID# 209997, Goyang, Gyeonggido
  - SoonChunHyang University Buchon Hospital /ID# 210618, Habun, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 210616, Seongnam, Gyeonggido
  - The Catholic University of Korea, ST. Vincent's Hospital /ID# 216951, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 209995, Suwon, Gyeonggido
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital /ID# 216949, Uijeongbu-si, Gyeonggido
  - Pusan National University Yangsan Hospital /ID# 214960, Yangsan, Gyeongsangnam-do
  - Wonkwang University Hospital /Id# 210620, Iksan, Jeonrabugdo
  - Kwangju Christian Hospital /ID# 210623, Gwangju, Jeonranamdo
  - Yonsei University Health System Severance Hospital /ID# 209636, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 210610, Seoul, Seoul Teugbyeolsi
  - Dongnam Institute of Radiological & Medical Sciences /ID# 209991, Busan
  - Good Samsun Hospital /ID# 209291, Busan
  - Inje University Busan Paik Hospital /ID# 209992, Busan
  - Inje University Haeundae Hospital /ID# 209993, Busan
  - Maryknoll Medical Center /ID# 210957, Busan
  - Dong-A University Hospital /ID# 209450, Busan
  - Pusan National University Hospital /ID# 209813, Busan
  - Kosin University Gospel Hospital /ID# 210608, Busan
  - Samsung Changwon Hospital /ID# 211507, Changwon
  - Samsung Changwon Hospital /ID# 211743, Changwon
  - Dankook University Hospital /ID# 209297, Cheonan
  - Chuncheon Sacred Heart Hospital /ID# 210612, Chuncheon
  - Kyungpook National University Chilgok Hospital /ID# 209988, Daegu
  - Keimyung University Dongsan Medical Center /ID# 212144, Daegu
  - Keimyung University Dongsan Medical Center /ID# 212514, Daegu
  - Kyungpook National University Hospital /ID# 209294, Daegu
  - Yeungnam University Medical Center /ID# 209293, Daegu
  - Kim Jun Hwan Sok Internal Medi /ID# 209292, Daegu
  - The Catholic University of Korea, Daejeon St.Mary's Hospital /ID# 216952, Daejeon
  - Chungnam National University Hospital /ID# 209637, Daejeon
  - Myongji Hospital /ID# 215595, Goyang
  - CHA Gumi Medical Center, CHA University /ID# 209994, Gumi
  - Chosun University Hospital /ID# 210607, Gwangju
  - The Catholic University of Korea Incheon St.Mary's Hospital /ID# 216950, Incheon
  - Gachon University Gil Medical Center /ID# 212513, Incheon
  - Inha University Hospital /ID# 210617, Incheon
  - Jeju National University Hospital /ID# 214700, Jeju City
  - Chonnam National University Hwasun Hospital /ID# 209990, Jeonnam
  - Inje University Sanggye Paik Hospital /ID# 210811, Seoul
  - Korea University Anam Hospital /ID# 210958, Seoul
  - Seoul National University Hospital /ID# 210959, Seoul
  - Seoul National University Hospital /ID# 211365, Seoul
  - Seoul National University Hospital /ID# 211369, Seoul
  - National Medical Center /ID# 209911, Seoul
  - Kangdong Sacred Heart Hospital /ID# 210621, Seoul
  - Asan Medical Center /ID# 210622, Seoul
  - Gangnam Severance Hospital /ID# 212512, Seoul
  - Samsung Medical Center /ID# 209296, Seoul
  - Samsung Medical Center /ID# 209635, Seoul
  - Chung-Ang University Hostipal /ID# 209295, Seoul
  - Ewha Womans University Mokdong Hospital /ID# 214961, Seoul
  - Ewha Womans University Mokdong Hospital /ID# 216412, Seoul
  - Korea University Guro Hospital /ID# 209989, Seoul
  - St. Carollo General Hospital /ID# 210619, Suncheon
  - Ulsan University Hospital /ID# 210810, Ulsan
  - Wonju Severance Christian Hospital /ID# 210611, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P19-423#additional-resources-section